CLINICAL TRIAL: NCT04111861
Title: Singing for Chronic Pain, a Pilot Study of a New Intervention for the Management of Chronic Pain
Brief Title: Singing for Chronic Pain, a New Intervention for the Management of Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019 RCHT 61
Record Dates: First submitted 2019-09-10; First posted 2019-10-01 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Singing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intevention (Experimental): To see if singing can be used as a detractive method from patients experiencing ongoing pain.
  Interventions: Other: Singing

INTERVENTIONS:
Other: Singing — To investigate whether singing can help people to manage their chronic pain the applicants, working together with people with chronic pain, have developed a singing intervention, Singing for Chronic Pain (SCP). The development of the programme has been supported by Snape Moultings, an international centre for the arts which offered the team a residency to develop the programme (https://snapemaltings.co.uk/music/residencies/). The model takes a holistic approach using voice and singing, movement, sound, mindfulness and breath work to provide opportunities to connect body, voice, breath and mind. This is important given that people often use body dissociation as a way to cope with physical pain

SUMMARY:
The aim of the project is to determine the feasibility of delivering a Singing for Chronic Pain (SCP) programme to patients with chronic pain attending a pain clinic.

The investigator will also be looking to provide a preliminary estimate of the benefit of SCP on self-efficacy, self -management skills, mindfulness and well-being as measured by standardized outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older and have a diagnosis of chronic pain with a duration of 6 months or more.

Exclusion Criteria:

* Having a mental health and/or physical health diagnosis that might prevent active engagement/participation in group sessions; Severe hearing impairment; Severe/profound cognitive impairment that may limit active engagement/participation in group sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-08-18 (Estimated); Study Completion 2022-08-18 (Estimated)

PRIMARY OUTCOMES:
Completion rate | One year
  Measure of attendance at sessions
Consent rate | One year
  Measure of those offered the programme who consent to take part

SECONDARY OUTCOMES:
Self reported self efficacy | One year
  Pain Self-efficacy questionnaire
Self reported ability to self-manage pain | One year
  Patient Activation Measure questionnaire
Increased mindfulness Increased mindfulness Increased mindfulness | One year
  Frieburg Mindfulness questionnaire
Self reported well-being | One year
  Edinburgh Warwick Well-being questionnaire
Self reported anxiety depression | One year
  Hospital Anxiety and Depression questionnaire.The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Anxiety scores and depression scores can range for 0 -21 with a higher score being worse. The separate depression and anxiety scores scores can be combined to give an overall score.
Self reported quality of life | One year
  EQ5D Quality of Life Questionnaire The EQ-5D questionnaire has two components: health state description and evaluation.Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondents self-rate their level of severity for each dimension using three-level (EQ-5D-3L) or five-level (EQ-5D-5L) scale.
  In the evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS).he answers given to ED-5D permit to find 243 unique health states or can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).

OTHER OUTCOMES:
Patient Focus Group | One year
  At week 10, participants will be invited to take part in a 60 minute focus group led by an experienced researcher. The focus groups will explore participants' perception of the programme and its outcomes, reasons for noncompliance, instrument appropriateness and suggestions for programme improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Cornwall Hospital, Truro, Cornwall, United Kingdom